CLINICAL TRIAL: NCT01183637
Title: Initial Safety and Effectiveness Study of the Kensey Nash Corp. Cartilage Repair Device for Knee Cartilage Lesion Repair
Brief Title: Evaluation of an Acellular Osteochondral Graft for Cartilage LEsions Pilot Trial
Acronym: EAGLE Pilot
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study enrollment rate was far slower than anticipated. Study was stopped for business purposes.
Sponsor: Kensey Nash Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EAGLE Pilot
Record Dates: First submitted 2010-07-28; First posted 2010-08-17 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Articular Cartilage Injury
Keywords: Cartilage; Knee; Osteochondral
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Patients assigned to the treatment arm will receive treatment with the Kensey Nash Corp. Cartilage Repair Device.
  Interventions: Device: Kensey Nash Corp. Cartilage Repair Device
- Control (Active Comparator): Patients assigned to the Control Arm will receive treatment with the standard surgical technique known as microfracture.
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Device: Kensey Nash Corp. Cartilage Repair Device — To perform the Cartilage Repair Device implantation procedure, the surgeon first removes the damaged cartilage. Then, the surgeon creates a cylindrical hole in the bone below the area of damaged cartilage. The Cartilage Repair Device is then implanted into the hole so that the surface is level with the surrounding native cartilage. The Cartilage Repair Device will then absorb blood and bone marrow from the bone to begin the healing process.
  Arms: Treatment
Procedure: Microfracture — To perform the microfracture technique, the surgeon will first remove the damaged cartilage. Then, the surgeon will make a number of small fractures in the bone below the area of damaged cartilage. The fractures cause the bone to bleed and a clot to form over the exposed bone. Over time, the clot forms a layer of fibrocartilage over the bone.
  Arms: Control

SUMMARY:
The Kensey Nash Corp. Cartilage Repair Device is a bioresorbable scaffold designed to promote repair of knee cartilage and subchondral bone. Subjects with knee cartilage damage meeting eligibility criteria will be randomly assigned to receive treatment with the Cartilage Repair Device or a standard surgical technique called microfracture. The purpose of the study is to evaluate the initial safety and effectiveness of the Cartilage Repair Device compared to microfracture.

DETAILED DESCRIPTION:
Damage to articular cartilage in the knee by acute or chronic injury causes pain and limits knee function. If left untreated, damage to the articular cartilage can lead to painful osteoarthritis. The human body has a limited ability to regenerate or adequately repair damage to articular cartilage. There are several surgical techniques available to assist the repair of articular cartilage and improve pain and function. Microfracture is the most commonly used technique for cartilage repair. Microfracture involves the creation of numerous small fractures in the bone with a pick. These small fractures cause the release of multipotential stem cells from the bone marrow creating a clot on the surface. Over time, this clot causes reparative fibrocartilage to form. However, fibrocartilage is less durable and lacks the mechanical properties of normal articular cartilage. The majority of patients treated with microfracture has good results within the first 2 years after microfracture. However, beyond 2 years, functional deterioration is seen in over 50% of patients. Therefore, there is a clinical need for a product that improves surgical outcomes in patients with cartilage damage.

The Kensey Nash Corp. Cartilage Repair Device is a two layer, bioresorbable implant. The top layer consists of collagen fibers like those found in normal cartilage. The collagen layer is about as thick as the cartilage in human knees. The bottom layer of the Cartilage Repair Device mainly consists of a calcium mineral naturally found in human bones. The mineral is held within a biodegradable polymer material. The device has a highly porous structure that allows the blood, stem cells and joint fluid to infiltrate the device during the healing process. Over time, the top layer is designed to be replaced by cartilage and the bottom layer is designed to be replaced by bone.

Both microfracture and the Cartilage Repair Device are expected to reduce knee pain and increase knee function in a majority of patients during the first 2 years post-operative. However, if the Cartilage Repair Device produces better and more durable cartilage than the microfracture technique, those patients treated with the Cartilage Repair Device may have a better long term outcome.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old and skeletally mature
* KOOS Pain subscale score is less than 65 (i.e. moderate pain)
* KOOS Activities of Daily Living score is less than 70 (i.e. moderate functional limitations)
* ICRS grade 3 or 4 cartilage lesion on the medial femoral condyle, lateral femoral condyle or trochlea measuring less than or equal to 15mm in diameter
* Stable meniscus with greater than 50% remaining bilaterally
* Mental capacity and willingness to comply with the post-operative rehabilitation plan and follow-up evaluations
* Written informed consent

Exclusion Criteria:

* Body mass index greater than 35
* Contraindication for MRI
* Previous microfracture, autograft implantation, allograft implantation or autologous chondrocyte implantation procedure on the damaged cartilage surface
* Knee ligament surgery within the past 6 months
* Clinically significant knee malalignment
* Osteoarthritis in the knee
* Multiple cartilage lesions
* Inflammatory arthropathy (i.e. rheumatoid arthritis, systemic lupus or active gout)
* Active infection in either lower limb
* Hyaluronic acid or cortisone injections within the past 3 months
* History of substance abuse
* Current participation in a study of an investigational product for a similar purpose
* Active litigation for the knee injury

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Patient Success | 24 months
  Improvement in pain, function, and cartilage defect appearance without any treatment related serious adverse events.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritic Outcome Score ("KOOS") | 24 months
  Clinically significant improvement in the KOOS Pain, Activities of Daily Living, Symptoms, Sports & Recreation and Quality of Life subscale scores
Cartilage defect appearance on MRI | 24 months
  Cartilage defect filling, repair cartilage integration with surrounding native cartilage and presence of bony overgrowth will be assessed.
Lyshom Score | 24 months
  Clinical significant improvement in the Lysolm Knee Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Lehman, M.D., Principal Investigator — U.S. Center for Sports Medicine, Kirkwood, MO; Phillip A Davidson, M.D., Principal Investigator — Heiden - Davidson Orthopedics, Park City, UT
Locations (2):
- United States (2):
  - Peninsula Orthopedic Associates, Salisbury, Maryland
  - U.S. Center for Sports Medicine, Kirkwood, Missouri